CLINICAL TRIAL: NCT03287505
Title: Evaluation of Pharmacokinetics and Safety of Aripiprazole IM Depot Formulation by Single Administration in Chinese Patients With Schizophrenia: a Single-center, Uncontrolled, Open -Label Trial
Brief Title: Aripiprazole IM Depot for Chinese Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 031-403-00050
Record Dates: First submitted 2017-05-15; First posted 2017-09-19 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abilify IM Depot 300mg by once (Experimental): 300 mg dose group: single-administration of Aripiprazole IM Depot (300 mg) in 12 subjects;
  Interventions: Drug: Aripiprazole IM Depot
- Abilify IM Depot 400mg by once (Experimental): 400 mg dose group: single-administration of Aripiprazole IM Depot (400 mg) in 12 subjects.
  Interventions: Drug: Aripiprazole IM Depot

INTERVENTIONS:
Drug: Aripiprazole IM Depot — administration of Aripiprazole IM Depot formulation at doses of 300 and 400mg once in patients with schizophrenia.
  Other Names: ABILIFY MAINTENA

SUMMARY:
This study assess pharmacokinetics and safety of single-administration of Aripiprazole IM Depot formulation at doses of 300 and 400mg in patients with schizophrenia.

DETAILED DESCRIPTION:
In this study, a single-center, single-dose, single-administration trial will be carried out in patients with schizophrenia diagnosed pursuant to The Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR), to evaluate pharmacokinetics and safety of single-administration aripiprazole IM Depot (300/400 mg) after its administration in 24 patients with oral tolerance of this drug.

In this study, the washout period before administration is designed as a 35-day duration before administration of the investigational drug (aripiprazoleIM Depot), screening period a 4-week duration (28 days) before administration of the investigational drug, observation period after administration a 20-week duration after administration of the investigational drug and hospital stay a minimum 35-day duration after administration of the investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, and their legal representatives(or their guardian ), who have signed the informed consent form(ICF);
2. Patients with a diagnosis of schizophrenia as defined by DSM-IV-TR (295.30, 295.10, 295.20,295.90 , 295.60);
3. subjects, both male and female, who are at age between 18 and 64 (also including 18 and 64 years of age) at time of informed consent.

Exclusion Criteria:

1. Patients who have other psychiatric disorders than schizophrenia based on diagnostic criteria of DSM-IV-TR;
2. Score of Positive and Negative Syndrome Scale (PANSS): ≥120;
3. Patients with a complication or a history of diabetic mellitus;
4. Subjects who are alcoholemia overdependent of drug, or have drug abuse history;

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | up to 20 weeks
  To assess the maximum Plasma Concentration (Cmax) of aripiprazole and its main metabolite OPC-14857
Time of Maximum Concentration | up to 20 weeks
  To assess the time of Maximum Concentration (tmax) of aripiprazole and its main metabolite OPC-14857
AUC0-∞ | up to 20 weeks
  To assess the area under the curve for period of medication, from 0 till infinity (AUC0-∞) of aripiprazole and its main metabolite OPC-14857
Apparent clearance after extravascular administration | up to 20 weeks
  To assess the Apparent clearance after extravascular administration (CL/F) of aripiprazole

SECONDARY OUTCOMES:
Adverse Events | up to 20 weeks
  Adverse events will be examined by frequency, severity, seriousness, discontinuation, and relationship to treatment.
Vital Signs | up to 20 weeks
  Mean change from baseline and the incidence of potentially clinically relevant abnormal values will be calculated for vital signs
Laboratory Examination | up to 20 weeks
  Mean change from baseline and the incidence of potentially clinically relevant abnormal values will be calculated for routine laboratory tests (including prolactin).

OTHER OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) | up to 20 weeks
  To evaluate the change of Positive and Negative Symptoms Scale (PANSS) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Master, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong F, Wang F, Yuan X, Zhai Y, Uki M, Jiang T, Li A. Single- and multiple-dose pharmacokinetics, safety, and tolerability of Aripiprazole once-monthly, long-acting intramuscular injection for Chinese adults with schizophrenia. BMC Psychiatry. 2025 Oct 1;25(1):912. doi: 10.1186/s12888-025-07407-w. PMID 41034820